CLINICAL TRIAL: NCT01711606
Title: EXPLAIN - FragilE X Registry: An exPlorative Longitudinal Study for chAracterIzation, Treatment Pathways and patieNt-related Outcomes
Brief Title: EXPLAIN -FragilE X Registry: An exPlorative Longitudinal Study for chAracterIzation, Treatment Pathways and patieNt-related Outcomes
Acronym: EXPLAIN
Status: Terminated | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAFQ056BDE-EPI-01
Record Dates: First submitted 2012-10-18; First posted 2012-10-22 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Fragile-X Syndrome
Keywords: Fragile-X Syndrome; registry; non-interventional trial; patient-related outcome study; drug utilization; effectiveness; treatment patterns; patient characteristics under real life conditions; quality of life; economics
MeSH Terms: conditions — Fragile X Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- unselected Fragile-X patients

SUMMARY:
This prospective observational study (registry) on Fragile X syndrome (FXS) is designed to evaluate characteristics, management and patient and caregiver-related outcomes the quality of life of Families and patients with FXS and to collect epidemiological and health economic data.

* EXPLAIN will report current and comprehensive data onEpidemiology data on fragile X syndrome
* Characterisation of the phenotype of FXS patients
* Description of patient characteristics (demographics, family history, comorbidity, education, working situations, care situations, insurance status)
* Documentation of therapeutic interventions
* Recording and assessment of psychosocial parameters (possibly also inclusion of family members, carers)
* quality of life of the carer and if possible the patient
* Health economic parameters and consumption of resources

ELIGIBILITY:
Inclusion Criteria:

* Patients with FXS as confirmed by genetic testing

Exclusion Criteria:

* none
* Other protocol-defined inclusion/exclusion criteria may apply

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with fragile-X Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2013-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Patient characteristics (demographics, family history, comorbidities, education, working situation, care situation, insurance status) | 3 years

SECONDARY OUTCOMES:
Epidemiology data on Fragile X Syndrome (FXS) | 3 years
Health-economic parameters and consumption of resources | 3 years
Therapeutic interventions and their application rationale | 3 Years
Psychosocial parameters (poss. also inclusion of family members, caregivers) | 3 years
Quality of life of the caregiver and possibly the patient | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Frank Hässler, MD, Principal Investigator — Klinik für Psychiatrie, Neurologie, Psychosomatik und Psychotherapie im Kindes- und Jugendalter, Gehlsheimer Straße 20, D- 18147 Rostock
Locations (1):
- Novartis Investigative site, Nuremberg, Germany

REFERENCES:
- [Derived] Haessler F, Gaese F, Huss M, Kretschmar C, Brinkman M, Peters H, Elstner S, Colla M, Pittrow D. Characterization, treatment patterns, and patient-related outcomes of patients with Fragile X syndrome in Germany: final results of the observational EXPLAIN-FXS study. BMC Psychiatry. 2016 Sep 10;16(1):318. doi: 10.1186/s12888-016-1020-5. PMID 27612457
- [Derived] Haessler F, Gaese F, Colla M, Huss M, Kretschmar C, Brinkman M, Schieb H, Peters H, Elstner S, Pittrow D. EXPLAIN Fragile-X: an explorative, longitudinal study on the characterization, treatment pathways, and patient-related outcomes of Fragile X Syndrome. BMC Psychiatry. 2013 Dec 19;13:339. doi: 10.1186/1471-244X-13-339. PMID 24354947